CLINICAL TRIAL: NCT00588822
Title: A Phase II Trial of Rituximab for Peripheral Neuropathy Associated With Monoclonal Gammopathy of Undetermined Significance (MGUS)
Brief Title: Rituximab in Treating Patients With Peripheral Neuropathy Caused by Monoclonal Gammopathy of Undetermined Significance
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Discontinuation due to the high response rate at the 1st stage and slow accrual.
Sponsor: Mayo Clinic (Other)
Collaborators: Genentech, Inc. (Industry); Biogen (Industry); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Alvaro Moreno Aspitia, Mayo Clinic - Jacksonville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1191-04; UL1RR024150 (NIH)
Record Dates: First submitted 2007-12-20; First posted 2008-01-09 (Estimated); Results first posted 2014-05-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-04

CONDITIONS: Precancerous Condition
Keywords: monoclonal gammopathy of undetermined significance
MeSH Terms: conditions — Precancerous Conditions; Monoclonal Gammopathy of Undetermined Significance | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab (Experimental): Subjects will receive rituximab administered at the standard dose and schedule as an initial cycle of therapy, followed by a re-evaluation at 6 months. If the neuropathy is stable or responding at 6 months, the subject will receive Cycle 2 of rituximab, followed by a re-evaluation at 12 months.
  Rituximab will be given as a 375 mg/m^2 intravenous infusion once weekly for four doses (days 1, 8, 15, and 22).
  Interventions: Biological: Rituximab

INTERVENTIONS:
Biological: Rituximab — Rituximab will be given as a 375 mg/m^2 intravenous infusion once weekly for four doses (days 1, 8, 15, and 22).
  Other Names: Rituxan

SUMMARY:
This study was done to find out if the investigational medication, rituximab, could help relieve the symptoms of peripheral neuropathy (such as numbness [abnormal protein in the blood] and weakness of the lower and upper extremities) in people who have monoclonal gammopathy of undetermined significance and people with a symptomatic or smoldering Waldestrom macroglobulinemia.

Rituximab is an antibody which attacks a particular type of white blood cell (B Cell). By targeting the B-cells which make the abnormal protein which is involved in causing the nerve trouble, it is hoped that damage to nerve fibers will be stopped and improvement will be allowed to proceed.

DETAILED DESCRIPTION:
This was a Phase II single arm trial evaluating the use of Rituximab administered at standard dose and schedule as an initial cycle of therapy, followed by a re-evaluation at 6 months.

If progression in neuropathy (as indicated by an increase in the Neuropathy Impairment Score (NIS) of greater than or equal to 10 or a modified Rankin Score increase of > 1 grade) the patient was off study. In addition, if the subject elected to pursue other active treatment including but not limited to plasmapheresis, high-dose intravenous immuneglobulin (IVIG), chemotherapeutic agents, or high dose corticosteroids, or if conditions in the exclusion criteria develop subsequent to enrollment, the subject was off study.

If the neuropathy is stable or responding (NIS of < 10 or a modified Rankin Score increase of < 1 grade) the patient would have received Cycle 2 of rituximab followed by a reevaluation at 12 months.

The study had a Simon Optimal two-stage Phase II design (α 5%, β 10%, π0 5%, π1 20%). The minimum clinically important response rate was 20%. The first stage was to include 21 patients and the second stage a total of 41 patients. The treatment would be rejected if there were fewer than 2 responders at the first stage or fewer than 5 responders at the second stage. The treatment would be accepted for further study if there were at least 5 responders out of 41 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of monoclonal gammopathy of undetermined significance (MGUS), as evidenced by 1 of the following criteria:

  * Documented monoclonal protein in the serum (< 3 g/dL) or urine
  * Monoclonal serum free light chain, with at least 50% of patients having an immunoglobulin M (IgM) paraprotein (the balance being immunoglobulin G (IgG) or immunoglobulin A (IgA) subtypes)
* Neuropathy Impairment Score (NIS) ≥ 25
* Stable or progressive neuropathy (i.e., not currently improving), as judged by NIS values that have not fallen ≥ 10 (between enrollment and the last documented value), at least 1 month but not greater than 3 months prior to enrollment
* No evidence of amyloidosis or overt lymphoma, overt myeloma, or Waldenström macroglobulinemia with end organ damage
* No evidence of multiple myeloma, Amyloid Light-chain (AL)-amyloidosis
* No evidence of Polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome, diabetes mellitus, alcohol induced neuropathy, untreated hypothyroidism, vitamin B12 deficiency, Sjögren syndrome, and other causes of neuropathy

PATIENT CHARACTERISTICS:

Inclusion Criteria:

* Not pregnant
* Negative serum pregnancy test
* Fertile patients must use an acceptable method of birth control during treatment and for 6 months after completion of treatment

  * One of the following birth control measures must be used: birth control pills, intrauterine device, contraceptive injections (Depo-Provera), barrier methods such diaphragm, condom or contraceptive sponge with spermicide
* Adequate bone marrow function as indicated by sufficient precursors of all three cell lines and cellularity of at least 20% on bone marrow biopsy within 6 months
* Platelets > 100,000/mm^3
* Absolute neutrophil count (ANC) > 1,000/mm^3
* Hemoglobin > 7 g/dL
* Serum creatinine < 3.0 mg/dL
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 2 times upper limit of normal
* No history of psychiatric disorder requiring hospitalization, psychiatric consultation, or psychotropic medications within the last year

  * Patients with controlled depression are eligible, as defined by the following:

    * Stable for at least 6 months
    * No increase in psychotropic medications

Exclusion criteria:

* History of HIV infection or seropositivity
* History or serological profile suggesting prior hepatitis B virus (HBV) infection (i.e., HbsAg or anti-HBs with anti-HBc)

  * Prior HBV vaccination with isolated anti-HBs antibodies is not an exclusion criterion
* HBV infection or non-vaccination-related HBV seropositivity
* Active infection
* New York Heart Association class III or IV heart disease
* History or baseline ECG tracing demonstrating severe recurrent or severe recent (within 3 months) cardiac dysrhythmia (e.g., ventricular tachycardia, torsades de pointes ("Twisting of the Points," a rapid polymorphic Ventricular Tachycardia), or other serious ventricular dysrhythmias) requiring implanted defibrillator treatment
* Confirmed diagnosis of systemic lupus erythematosus (SLE)

  * An isolated low titer positive antinuclear antibody test without clinical evidence of SLE is not an exclusion criterion
* Concomitant malignancies or previous malignancies within the last five years, with the exception of adequately treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Malignancy associated with a paraneoplastic neuropathy
* A history of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* A history of known severe primary or secondary immunodeficiency (e.g., common variable immunodeficiency)
* Significant other uncontrolled medical illnesses that may interfere with drug delivery or interpretation of results

PRIOR CONCURRENT THERAPY:

* No live vaccine therapy within 30 days of enrollment
* No plasmapheresis within 3 months
* No high-dose intravenous immunoglobulin, chemotherapeutic agents, or high-dose corticosteroids (> 10 mg daily or every other day) within 3 months
* No systemic corticosteroids within 3 months (unless needed for adrenal insufficiency or at a stable dose ≤ 10 mg daily)
* No high-dose (> 250 mg/day) vitamin B6 within the past month
* No prior treatment with thalidomide or neurotoxic drugs (e.g., vinca alkaloids, taxol, or platinum)

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-01; Primary Completion 2009-01 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benn E. Smith, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Mayo Clinic Cancer Center, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enroll from January 2005 to June 2008 at the Mayo Clinic in Arizona, Florida, and Minnesota.
Period: Overall Study
Arm/Group | Rituximab
Started | 21
Completed | 13
Not Completed | 8
Not completed — progression of disease | 8

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With at Least 10 Points Improvement in the Neuropathy Impairment Score (NIS) for Either Side of the Body at 6 Months
Description: The Neuropathy Impairment Score [previously called the Neurologic Disability Score (NDS)] is derived from a neurologic examination obtained in a standard way by a specially trained neurologist. Decisions are based on the neurologist's judgment of what is normal considering site, age, sex, weight, height, and physical fitness. The instrument has 35 items, each ranked for left and right sides of the body; weakness is scored 0=normal, 1=25% disability, 2=50% disability, 3=75% disability and 4=100% disability. NIS total score was calculated as the sum of the 35 items, ranging from 0 to 140, with higher score indicating greater disability or impairment.
  The neurologist measured the NIS score on both sides of the body, but recorded worst score and reported as 1 for each individual subject (i.e., each subject had only 1 reported score.)
  Improvement was defined as at least 10 points improvement in NIS total score, that is, reduction in the number of points on the scale.
Time Frame: baseline, 6 months
Population: A dichotomous measure was used so that subjects who discontinued participation prematurely could be included as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Rituximab
Number analyzed (Participants) | 21
percentage of subjects | 62 [38 to 82]

2. Secondary Outcome: Percentage of Subjects Whose Disease Has Stabilized or Responded, for Either Side of the Body, as Measured by NIS at 6 Months
Description: The Neuropathy Impairment Score (previously called the Neurologic Disability Score [NDS]) is derived from a neurologic examination obtained in a standard way by a specially trained neurologist. Decisions are based on the neurologist's judgment of what is normal considering site, age, sex, weight, height, and physical fitness. The instrument has 35 items, each ranked for left and right sides of the body; weakness is scored 0=normal, 1=25% disability, 2=50% disability, 3=75% disability and 4=100% disability. NIS total score was calculated as the sum of the 35 items, ranging from 0 to 140, with higher score indicating greater disability or impairment.
  The NIS score was measured on both sides of the body, the worst score recorded reported as 1 for each individual subject. Stability was defined as change of less than 10 points in the NIS total score. Improvement was defined as at least 10 points improvement in NIS total score, that is, reduction in the number of points on the scale.
Time Frame: baseline, 6 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Rituximab
Number analyzed (Participants) | 21
percentage of subjects | 86 [64 to 97]

3. Secondary Outcome: Percentage of Subjects With at Least 1 Grade Improvement in the Modified Rankin Score at 6 Months
Description: The Modified Rankin Scale was used to determine functional disability as follows: 0 = asymptomatic; 1 = symptoms not interfering with manual activities/walking normally; 2 = minor difficulties in manual activities/walking independently without support; 3 = unable to perform some manual activities/walking independently with support; 4 = unable to eat, dress or wash independently/needing assistance to walk; 5 = no useful tasks performed with upper limbs/confined to wheelchair. Therefore, scores could range from 0 to 5, with higher values indicating greater disability.
Time Frame: baseline, 6 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Rituximab
Number analyzed (Participants) | 21
percentage of subjects | 19 [5 to 42]

4. Secondary Outcome: Percentage of Patients Having Improvement in the Hand Grip Strength Ergometry Value for Either Hand at 6 Months
Description: Grip strength was measured by a dynamometer in both hands at baseline and every three months until the final study visit. Response criteria was defined as achieving improvement in hand grip strength dynamometry values (>10% better relative to baseline at the 6 month visit on either side).
Time Frame: baseline, 6 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Rituximab
Number analyzed (Participants) | 21
percentage of subjects | 52 [30 to 74]

5. Secondary Outcome: Percentage of Subjects Having One or More Stable Hand Grip Strength Ergometry Values for Either Hand at 6 Months
Description: Grip strength was measured by a dynamometer in both hands at baseline and every three months until the final study visit. Response criteria was defined as achieving stable hand grip strength dynamometry values (no more than 10% better or worse relative to baseline at the 6 month visit on either side).
Time Frame: baseline, 6 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Rituximab
Number analyzed (Participants) | 21
percentage of subjects | 76 [53 to 92]

6. Secondary Outcome: Percentage of Subjects With > 50% Reduction of Monoclonal Protein Titer at 6 Months
Description: Monoclonal immunoglobulins measured included Immunoglobulin G (IgG), Immunoglobulin A (IgA), and Immunoglobulin M (IgM).
Time Frame: baseline, 6 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Rituximab
Number analyzed (Participants) | 21
percentage of subjects
  IgG Responder | 0 [0 to 17]
  IgA Responder | 0 [0 to 17]
  IgM Responder | 5 [0 to 25]

ADVERSE EVENTS:
Time Frame: Subjects were monitored for adverse events weekly per cycle ( Day 1, 8, 15, and 22); each subject could receive up to 2 cycles (4 infusions each.) Adverse event monitoring continued for at least 12 months following the subject's last Rituximab infusion.
Arm/Group | Rituximab
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=21)
Myocardial infarction (Cardiac disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was discontinued at the first stage to the high response rate and slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No